CLINICAL TRIAL: NCT06663956
Title: A Randomized Controlled, Open Clinical Trial of a Web-based Platform for Multifactorial Intervention in Cancer Pain Management
Brief Title: A Randomized Controlled Trial of a Web-based Platform for Cancer Pain Management
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, PhD, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-1948
Record Dates: First submitted 2024-10-26; First posted 2024-10-29 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Cancer Pain
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The conventional treatment paradigm is in the current paradigm of standard antitumor cancer pain treatment and follow-up with no warning and no patient feedback.
- Experimental group (Experimental): We propose to develop a patient self-reporting applet that is easy to use and simple to operate. The program is embedded with questionnaires related to cancer pain and quality of life assessment, so that patients can fill out the questionnaires to report their symptoms and changes in their conditions to primary care doctors in a timely manner. At the same time, the background of the program will monitor the patient's indicators in real time. When the patient's pain reaches moderate-to-severe level, or when the patient experiences side effects of drugs, or when the patient's adherence to medication is poor, the primary care doctor can immediately receive relevant alerts through the app, so as to intervene in the patient's cancer pain treatment. When the patient has an "alarm value", primary care doctors can provide feedback to doctors in higher-level hospitals and implement comprehensive and standardized treatment for cancer pain patients.
  Interventions: Behavioral: a patient self-reporting applet

INTERVENTIONS:
Behavioral: a patient self-reporting applet — We propose to develop a patient self-reporting applet that is easy to use and simple to operate. The program is embedded with questionnaires related to cancer pain and quality of life assessment, so that patients can fill out the questionnaires to report their symptoms and changes in their conditions to primary care doctors in a timely manner. At the same time, the background of the program will monitor the patient's indicators in real time. When the patient's pain reaches moderate-to-severe level, or when the patient experiences side effects of drugs, or when the patient's adherence to medication is poor, the primary care doctor can immediately receive relevant alerts through the app, so as to intervene in the patient's cancer pain treatment. When the patient has an "alarm value", primary care doctors can provide feedback to doctors in higher-level hospitals and implement comprehensive and standardized treatment for cancer pain patients.
  Arms: Experimental group

SUMMARY:
Malignant tumors are one of the major public health problems in China, and cancer pain is a common symptom in tumor patients, affecting the quality of life. In rural areas, cancer pain management is challenging due to insufficient medical resources and limitations in understanding cancer pain. Investigators plan to develop a convenient patient self-reporting applet to help participants report their symptoms to primary care physicians promptly and monitor pain levels and medication in real-time. This project aims to improve the efficiency of cancer pain management, integrate cancer pain into chronic disease management, improve the quality of healthcare services for rural participants, and promote the construction of a healthy China.

ELIGIBILITY:
Inclusion Criteria:

* Patients with tumors that are confirmed by pathological findings.
* Presence of tumor-related pain that is moderate or higher and requires intervention with morphine-based pain medication (++).
* Have a life expectancy of more than 6 months.
* Understand and sign a consent to participate in the study, or if the patient is unable to understand the study, his/her direct caregiver must have a good understanding of the study.

Exclusion Criteria:

* Presence of other chronic non-cancer pain/have an unresolved pain-related condition.
* Moderately severe cognitive impairment/cognitive impairment.
* Have schizophrenia or other psychiatric illness.
* Neither the patient nor his/her direct caregiver can understand how to use the Cancer Pain Management applet.
* Being pregnant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-10 (Actual); Primary Completion 2026-11-10 (Estimated); Study Completion 2026-11-10 (Estimated)

PRIMARY OUTCOMES:
Patient's average pain level (derived from the Brief Pain Scale) | From patient enrollment to 3 months, during which time the applet was used once a week
  The Brief Pain Inventory (BPI) is a validated tool for assessing pain intensity and impact on daily life.
  The BPI consists of two parts: the first part assesses the intensity of pain using a scale of 0 to 10, where 0 indicates no pain and 10 indicates the worst pain; the second part assesses the impact of pain on various aspects of the patient's life (e.g., mood, work, sleep, and social activities).
  The BPI is simple and easy to use, and can help healthcare professionals to quickly obtain quantitative information about pain and monitor the effectiveness of pain management.

SECONDARY OUTCOMES:
Mood and physical state of the patient (derived from the EQ-5D scale) | From patient enrollment to 3 months, during which time the applet was used twice a week
  The EQ-5D is a brief scale used to assess an individual's health status and quality of life.The EQ-5D provides a standardized assessment of a patient's health-related quality of life. The scale consists of two parts: the first part is a self-assessment of five dimensions, including mobility, self-care, activities of daily living, pain/discomfort, and anxiety/depression, each of which is scored on a scale ranging from "no problem," "mild problem," "moderate problem," "moderate problem," "moderate problem," "moderate problem," "moderate problem," "moderate problem," "moderate problem," "moderate problem," "moderate problem," and "moderate problem, "Moderate Problems, Severe Problems, and Extreme Problems. The second part is a visual analog scale (VAS) that assesses general health on a scale from 0 (very poor health) to 100 (optimal health).
Burden situation of family members (derived from the Family Support Scale) | From patient enrollment to 3 months, during which time the applet was used twice a week
  The Family Support Scale (FSS) is an instrument used to assess the level of support an individual receives in their home environment. The Family Support Scale usually contains items along multiple dimensions, such as emotional support (e.g., care and understanding), material support (e.g., material help), informational support (e.g., advice and guidance), and other relevant family interaction factors. Respondents rate their feelings and experiences of family support, usually on a Likert scale, e.g., from "completely disagree" to "completely agree."
Patient quality of life (derived from the QLQ-C30 core quality of life questionnaire) | From patient enrollment to 3 months, during which time the applet was used twice a week
  The C30 scale (EORTC QLQ-C30) is an instrument developed by the European Organization for Research and Treatment of Cancer (EORTC) to assess the quality of life of cancer patients. The scale consists of 30 entries covering the two main dimensions of functioning (e.g., physical, emotional, and social functioning) and symptoms (e.g., pain, fatigue), as well as general health. Patients are scored based on how they have felt over the past week, with scores typically ranging from 0 to 100. Higher scores indicate better quality of life, higher functional status, and less severe symptoms, while lower scores indicate poorer quality of life, limited functioning, and more severe symptoms.The C30 Scale is widely used in cancer research and clinical practice to monitor patients' health status and treatment outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan Universit, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No